CLINICAL TRIAL: NCT02163226
Title: A Randomized Trial Evaluating Rapid Delivery of Dose Escalated Hypofractionated Radiotherapy for Patients Diagnosed With Bone Metastases for Effective Palliation of Symptoms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0640; NCI-2014-01482 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-06-09; First posted 2014-06-13 (Estimated); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Bone Metastases
Keywords: Bone metastases; Hypofractionated Radiation Therapy; Standard Radiation Therapy; XRT; Pain control; Palliation of symptoms; Questionnaire; Survey
MeSH Terms: conditions — Agnosia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypofractionated Radiation Therapy (Experimental): Participants receive standard hypofractionated regimen of 3 Gy x 10 fractions, 1 radiation treatment a day for 5 days in a row. Questionnaire completion at months 1, 2, 3, 4, and 6 and then every 3 months after that for at least 3 years. Questionnaires ask about pain, pain relief, and quality of life.
  Interventions: Radiation: Hypofractionated Radiation Treatment; Behavioral: Questionnaire
- One Radiation Therapy Treatment (Active Comparator): 12 Gy x 1 fraction or 16 Gy x 1 fractions adaptively depending on the size of the metastases or gross tumor volume (GTV). Questionnaire completion at months 1, 2, 3, 4, and 6 and then every 3 months after that for at least 3 years. Questionnaires ask about pain, pain relief, and quality of life.
  Interventions: Radiation: One Radiation Treatment; Behavioral: Questionnaire

INTERVENTIONS:
Radiation: Hypofractionated Radiation Treatment — Participants receive standard hypofractionated regimen of 3 Gy x 10 fractions, 1 radiation treatment a day for 5 days in a row.
  Other Names: XRT
  Arms: Hypofractionated Radiation Therapy
Radiation: One Radiation Treatment — 12 Gy x 1 fraction or 16 Gy x 1 fractions adaptively depending on the size of the metastases or gross tumor volume (GTV).
  Other Names: XRT
  Arms: One Radiation Therapy Treatment
Behavioral: Questionnaire — Questionnaire completion at months 1, 2, 3, 4, and 6 and then every 3 months after that for at least 3 years. Questionnaires ask about pain, pain relief, and quality of life.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to learn if 1 large dose of radiation therapy is better at controlling pain from cancer that has spread to the bones than 10 smaller doses of radiation. Researchers also want to learn if 1 large dose of radiation therapy can help decrease the use of drugs to control the pain, and if it can help to control the disease.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group. You will have an equal chance of being assigned to either group.

If you are in Group 1, you will receive 1 radiation treatment a day for 10 days in a row (not counting weekends or holidays). You will receive a higher total dose of radiation than Group 2.

If you are in Group 2, you will receive 1 radiation treatment given on 1 day.

Radiation Therapy:

You will lie on a table for the radiation treatment(s). Each treatment will last about 30 minutes.

Length of Treatment:

You may receive 1 or 10 radiation treatments, depending on which group you are in. You will no longer be able to receive radiation therapy if intolerable side effects occur or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

Follow-Up Visits:

At Months 3, 6, 9, 12 and every 3 to 6 months after the start of radiation therapy, you will have x-rays, a bone scan, CT scan, or MRI to check the status of the disease.

At Months 3, 4, and 6 and then every 3 months after that for at least 3 years, you will complete the questionnaires about the pain, your pain relief, and your quality of life. The questionnaires can be filled out at a clinic visit or sent back in the mail.

This is an investigational study. Radiation therapy is delivered using FDA-approved and commercially available methods. It is investigational to compare the number and size of radiation doses.

Up to 300 participants will take part in this multicenter study. Up to 300 participants will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathologic diagnosis of malignancy
2. Patients with any radiographic evidence of bone metastases, including plain x-ray, bone scan, computed tomography (CT) scan, magnetic resonance imaging (MRI), or positron emission tomography (PET) scan
3. Patients with pain or dysaesthesia
4. Patients with a life expectancy of more than 3 months
5. Patients able to complete pain assessment and quality of life surveys
6. Patients with multiple osseous sites are eligible; however should not treat more than 3 separate radiation treatment fields concurrently.
7. Patients with surgery for osseous metastases are allowed.

Exclusion Criteria:

1. Patients with prior radiation therapy to the treatment site
2. Patients with a current, untreated spinal cord compression
3. Patients with a radiographic or pathologic fracture to the treatment site
4. Patients with painful metastases to hands and feet that need to be radiated on protocol
5. Patients previously treated with radioactive isotope (e.g. Sr89) within 30 days of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2014-08-06 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-nhu Nguyen, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - MD Anderson Cancer Center at Cooper, Voorhees Township, New Jersey
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Nguyen QN, Chun SG, Chow E, Komaki R, Liao Z, Zacharia R, Szeto BK, Welsh JW, Hahn SM, Fuller CD, Moon BS, Bird JE, Satcher R, Lin PP, Jeter M, O'Reilly MS, Lewis VO. Single-Fraction Stereotactic vs Conventional Multifraction Radiotherapy for Pain Relief in Patients With Predominantly Nonspine Bone Metastases: A Randomized Phase 2 Trial. JAMA Oncol. 2019 Jun 1;5(6):872-878. doi: 10.1001/jamaoncol.2019.0192. PMID 31021390
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There was total 167 patients enrolled in this phase II 2013-0640 palliation of symptoms study. Eligible criteria: pathologic diagnosis of malignancy; any radiographic evidence of bone metastases; with pain or dysathesia; life expectancy of more than 3 months; should not treat more than 3 separate radiation treatment fields concurrently.
Pre-assignment Details: A total of 167 patients were consented to this study, but 1 patient withdrew consent prior to protocol treatment, 3 patients insurance denied, 2 Patient condition deteriorated, 1 Pathologic fracture on reevaluation, only 160 patients was randomized and treated under this protocol.
Groups:
- Arm 1: the Standard Hypofractionated Regimen (MFRT Group): 3 Gy x 10 fractions; Patients can be treated with 2-D, 3-D, or intensity modulated radiation therapy (IMRT)
- Arm 2: Single-fraction Stereotactic Radiation (SBRT Group): 12 Gy x 1 fraction or 16 Gy x 1 fractions, depending on the size of the metastases or gross tumor volume (GTV), treated with 2-D, 3-D, or IMRT
Period: Overall Study
Arm/Group | Arm 1: the Standard Hypofractionated Regimen (MFRT Group) | Arm 2: Single-fraction Stereotactic Radiation (SBRT Group)
Started | 79 | 81
Completed | 63 | 70
Not Completed | 16 | 11
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Returned home, local radiotherapy | 3 | 0
Not completed — Repeat imaging showed no disease | 2 | 0
Not completed — Incomplete radiotherapy | 3 | 0
Not completed — Treatment was to >3 radiotherapy fields | 1 | 0
Not completed — "Insurance denied for single-fraction treatment" | 0 | 5
Not completed — ineligible | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: the Standard Hypofractionated Regimen (MFRT Group) | Arm 2: Single-fraction Stereotactic Radiation (SBRT Group) | Total
Number analyzed (Participants) | 79 | 81 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 36 | 76
  >=65 years | 39 | 45 | 84
Age, Continuous [Median (Full Range); unit: years] | 63 [23 to 84] | 63 [42 to 86] | 63 [23 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 47 | 49 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 69 | 73 | 142
  Unknown or Not Reported | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 2 | 10
  White | 59 | 68 | 127
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 79 | 81 | 160
Number of Lesions [Count of Participants; unit: Participants]
  ≤4 | 41 | 42 | 83
  >4 | 38 | 39 | 77
Site of Bony Mets [Count of Participants; unit: Participants]
  Abdomen | 4 | 3 | 7
  Thorax | 9 | 10 | 19
  Extremities | 13 | 15 | 28
  Head/Neck | 2 | 4 | 6
  Pelvis | 48 | 46 | 94
  Spine | 3 | 3 | 6
Numbers of Sites Irradiated [Count of Participants; unit: Participants]
  1 | 64 | 61 | 125
  >1 | 15 | 20 | 35
Karnofsky performance score (KPS) [Count of Participants; unit: Participants] — KPS 100: normal activity, 90: able to carry on normal activity, 80: normal activity with effort; 70: unable to carry on normal activity; 60: Requires occasional assistance, 50: Requires frequent assistance and medical care. The KPS was to allow physicians to evaluate a patient's survival. The higher KPS scores, the better treatment outcome.
  Participants
    KPS 50-60 | 10 | 9 | 19
    KPS 70-80 | 58 | 57 | 115
    KPS 90-100 | 11 | 15 | 26
Primary Cancer Site [Count of Participants; unit: Participants]
  Adrenal-cortical | 1 | 0 | 1
  Bladder | 4 | 3 | 7
  Breast | 3 | 11 | 14
  Esophagus | 4 | 4 | 8
  Head and Neck | 1 | 2 | 3
  Liver | 0 | 3 | 3
  Lung | 47 | 32 | 79
  Pancreas | 0 | 1 | 1
  Prostate | 9 | 14 | 23
  Renal Cell | 5 | 9 | 14
  Thymoma | 1 | 0 | 1
  Thyroid | 2 | 0 | 2
  Unknown/Lung | 0 | 1 | 1
  Uveal Melanoma | 1 | 0 | 1
  Multiple Myeloma | 1 | 1 | 2
Primary Tumor Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 50 | 51 | 101
  Adenoid Cystic | 1 | 0 | 1
  Adrenal Cortical Carcinoma | 1 | 0 | 1
  Atypical Carcinoid | 1 | 1 | 2
  Carcinoma | 1 | 1 | 2
  Clear Cell | 5 | 9 | 14
  Ductal Carcinoma | 0 | 4 | 4
  Lobular Carcinoma | 1 | 1 | 2
  Melanoma | 1 | 0 | 1
  Neuroendocrine | 1 | 3 | 4
  Papillary | 2 | 0 | 2
  Pleiomorphic Carcinoma | 1 | 0 | 1
  Poorly Diff Carcinoma | 1 | 0 | 1
  Sarcomatoid | 1 | 0 | 1
  Small Cell | 1 | 3 | 4
  Squamous | 6 | 5 | 11
  Urothelial Carcinoma | 4 | 4 | 8
  Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Intent- to- Treat Patients With Pain Response by Treatment
Description: Evaluate single fraction stereotactic regimen for pain response in terms of time to failure. Pain response was defined by international consensus criteria as a combination of pain score and analgesic use (daily morphine-equivalent dose). Pain failure (ie, lack of response) was defined as worsening pain score (2 points on a 0-to-10 scale), an increase in morphine-equivalent opioid dose of 50% or more, reirradiation, or pathologic fracture. Time to failure was defined as the first occurrence of any of the following events: worsening in pain score by at least 2 categories by MDASI survey. Statistical tests in treatment group were based on the Wilcoxon rank sum test to compare changes in pain scores and analgesic use at each assessment point relative to baseline. Increases or decreases of 2 or more points on a scale of 0 to 10 indicated improving or worsening pain. Fisher exact tests were used to compare the distribution of pain responders (CR + PR) and nonresponders (PP + IR).
Time Frame: From date of registration until the date of first documented Pain failure or death from any cause, or lost to follow up, whichever came first, assessed up to 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: the Standard Hypofractionated Regimen (MFRT Group) | Arm 2: Single-fraction Stereotactic Radiation (SBRT Group)
Number analyzed (Participants) | 79 | 81
Participants
  Pain Response (CR+PR) at 2 weeks | 19 | 34
  Pain Response (CR+PR) at 1 month | 24 | 36
  Pain Response (CR+PR) at 3 months | 17 | 31
  Pain Response (CR+PR) at 6 months | 17 | 19
  Pain Response (CR+PR) at 9 months | 12 | 17
Statistical Analysis 1: Comparison: Arm 1: the Standard Hypofractionated Regimen (MFRT Group); Pain Response Rates (CR+PR) at 2 weeks; Test type: Other — 2 sided p value; p = .03, Fisher Exact
Statistical Analysis 2: Comparison: Arm 1: the Standard Hypofractionated Regimen (MFRT Group) vs Arm 2: Single-fraction Stereotactic Radiation (SBRT Group); Pain Response Rates (CR+PR) at 1 month; Test type: Superiority; p = .19, Fisher Exact
Statistical Analysis 3: Comparison: Arm 1: the Standard Hypofractionated Regimen (MFRT Group); Pain Response Rates (CR+PR) at 3 months; Test type: Other — 2 sided p value; p = .04, Fisher Exact
Statistical Analysis 4: Comparison: Arm 1: the Standard Hypofractionated Regimen (MFRT Group); Pain Response Rates (CR+PR) at 6 months; Test type: Superiority; p = .89, Fisher Exact
Statistical Analysis 5: Comparison: Arm 1: the Standard Hypofractionated Regimen (MFRT Group); Pain Response Rates (CR+PR) at 9 months; Test type: Superiority; p = .07, Fisher Exact
Statistical Analysis 6: Comparison: Arm 2: Single-fraction Stereotactic Radiation (SBRT Group); Pain Response Rates (CR+PR) at 2 weeks; Test type: Other — 2 sided p value; p = .03, Fisher Exact
Statistical Analysis 7: Comparison: Arm 2: Single-fraction Stereotactic Radiation (SBRT Group); Pain Response Rates (CR+PR) at 1 month; Test type: Other — 2 sided p value; p = .19, Fisher Exact
Statistical Analysis 8: Comparison: Arm 2: Single-fraction Stereotactic Radiation (SBRT Group); Pain Response Rates (CR+PR) at 3 months; Test type: Other — 2 sided p value; p = .04, Fisher Exact
Statistical Analysis 9: Comparison: Arm 2: Single-fraction Stereotactic Radiation (SBRT Group); Pain Response Rates (CR+PR) at 6 months; Test type: Other — 2 sided p value; p = .89, Fisher Exact
Statistical Analysis 10: Comparison: Arm 2: Single-fraction Stereotactic Radiation (SBRT Group); Pain Response Rates (CR+PR) at 9 months; Test type: Other — 2 sided p value; p = .07, Fisher Exact

2. Primary Outcome: Number of Evaluable Participants With Pain Response by Treatment
Description: Evaluate single fraction stereotactic regimen for pain response in terms of time to failure. Pain response was defined by international consensus criteria as a combination of pain score and analgesic use (daily morphine-equivalent dose). Pain failure (ie, lack of response) was defined as worsening pain score (2 points on a 0-to-10 scale), an increase in morphine-equivalent opioid dose of 50% or more, reirradiation, or pathologic fracture. Time to failure was defined as the first occurrence of any of the following events: worsening in pain score by at least 2 categories by MDASI survey. Complete response (CR) is a pain score of 0 at the treated site and no increase in analgesic. Partial response (PR): reduction in pain score of 2 or more points above baseline with no increase in analgesic. Pain progression (PP): Increases of 2 or more points on a scale of 0 to 10 or worsening pain. indeterminate response (IR): were all other responses.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: the Standard Hypofractionated Regimen (MFRT Group) | Arm 2: Single-fraction Stereotactic Radiation (SBRT Group)
Number analyzed (Participants) | 52 | 55
Participants
  Pain Response (CR+PR) at 2 weeks | 19 | 34
  Pain Response (CR+PR) at 1 month | 24 | 36
  Pain Response (CR+PR) at 3 months | 17 | 32
  Pain Response (CR+PR) at 6 months | 17 | 19
  Pain Response (CR+PR) at 9 months | 12 | 17
Statistical Analysis 1: Comparison: Arm 1: the Standard Hypofractionated Regimen (MFRT Group); Pain response Rates (CR+PR) at 2 weeks; Test type: Other — 2 sided p value; p = .01, Fisher Exact
Statistical Analysis 2: Comparison: Arm 1: the Standard Hypofractionated Regimen (MFRT Group); Pain response Rates (CR+PR) at 1 month; Test type: Other — 2 sided p value; p = .15, Fisher Exact
Statistical Analysis 3: Comparison: Arm 1: the Standard Hypofractionated Regimen (MFRT Group); Pain response Rates (CR+PR) at 3 months; Test type: Other — 2 sided p value; p = .04, Fisher Exact
Statistical Analysis 4: Comparison: Arm 1: the Standard Hypofractionated Regimen (MFRT Group); Pain response Rates (CR+PR) at 6 months; Test type: Other — 2 sided p valued; p = .78, Fisher Exact
Statistical Analysis 5: Comparison: Arm 1: the Standard Hypofractionated Regimen (MFRT Group); Pain response Rates (CR+PR) at 9 months; Test type: Other — 2 sided p valued; p = .04, Fisher Exact
Statistical Analysis 6: Comparison: Arm 2: Single-fraction Stereotactic Radiation (SBRT Group); Pain response Rates (CR+PR) at 2 weeks; Test type: Other — 2 sided p valued; p = .01, Fisher Exact
Statistical Analysis 7: Comparison: Arm 2: Single-fraction Stereotactic Radiation (SBRT Group); Pain response Rates (CR+PR) at 1 month; Test type: Other — 2 sided p value; p = .15, Fisher Exact
Statistical Analysis 8: Comparison: Arm 2: Single-fraction Stereotactic Radiation (SBRT Group); Pain response Rates (CR+PR) at 3 months; Test type: Other — 2 sided p value; p = .04, Fisher Exact
Statistical Analysis 9: Comparison: Arm 2: Single-fraction Stereotactic Radiation (SBRT Group); Pain response Rates (CR+PR) at 6 months; Test type: Other — 2 sided p value; p = .78, Fisher Exact
Statistical Analysis 10: Comparison: Arm 2: Single-fraction Stereotactic Radiation (SBRT Group); Pain response Rates (CR+PR) at 9 months; Test type: Other — 2 sided p value; p = .04, Fisher Exact

3. Secondary Outcome: Number of Participants With Toxicity Associated With Treatment
Description: Report grade 3 acute (skin, fatigue, flare reaction) and long term (sclerosis, bone ossification, bone fracture rate) toxicity associated with treatment. During radiotherapy, the patient will be examined weekly and acute reactions recorded and toxicity occurring after 3 months of radiation therapy.
Time Frame: From date of registration until the date of documented death from any cause, or lost to follow up, whichever came first, assessed up to 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: the Standard Hypofractionated Regimen (MFRT Group) | Arm 2: Single-fraction Stereotactic Radiation (SBRT Group)
Number analyzed (Participants) | 79 | 81
Participants
  Nausea | 4 | 1
  Vomiting | 2 | 0
  Fatigue | 4 | 9
  Radiation Dermatitis | 2 | 1
  Fracture | 0 | 1

ADVERSE EVENTS:
Time Frame: From the time of registration to the time of the adverse events (AEs) start date, assessed up to 2 years
Arm/Group | Arm 1: the Standard Hypofractionated Regimen (MFRT Group) | Arm 2: Single-fraction Stereotactic Radiation (SBRT Group)
All-Cause Mortality (participants affected / at risk) | 49/79 | 42/81
Serious Adverse Events (participants affected / at risk) | 19/79 | 11/81
Other Adverse Events (participants affected / at risk) | 0/79 | 0/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: the Standard Hypofractionated Regimen (MFRT Group) (N=79) | Arm 2: Single-fraction Stereotactic Radiation (SBRT Group) (N=81)
Bone pain (Musculoskeletal and connective tissue disorders) | 15 (18) | 5 (6)
Fatigue (General disorders) | 4 (4) | 9 (9)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT02163226/Prot_SAP_000.pdf